CLINICAL TRIAL: NCT06739382
Title: Management of Ventilation Acquired Pneumonia Caused by Pseudomonas and Acinetobacter Organisms in a Pediatric Center: a Randomized Controlled Study
Brief Title: Management of Ventilation Acquired Pneumonia Caused by Pseudomonas and Acinetobacter Organisms in a Pediatric Center
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama, Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: code MS-280-2020
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Ventilation Acquired Pneumonia
Keywords: ventilator-associated pneumonia; pandrug-resistant; extensively drug-resistant
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Polymyxins; Tigecycline; Ertapenem; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- extended meropenem infusion in combination with other options (Active Comparator): a) Patients treatment was modified to extended meropenem infusion in combination with other options such as Polymyxin, Tigecycline, Ertapenem, or Amikacin
  Interventions: Combination Product: extended meropenem infusion in combination with other options such as Polymyxin, Tigecycline, Ertapenem, or Amikacin.
- two β-lactam antibiotics plus a single non-β-lactam antibiotic (Active Comparator): b) Patient treatment was adjusted to include two β-lactam antibiotics plus a single non-β-lactam antibiotic, or a combination of double β-lactam antibiotics, with the aim of avoiding aggressive and toxic antibiotics
  Interventions: Combination Product: two β-lactam antibiotics plus a single non-β-lactam antibiotic
- c) Patients treatment was adjusted to the second-line empirical antibiotic (Other): c) Control group in which patients treatment was adjusted to the second-line empirical anti-biotic according to the hospital's local policy.
  Interventions: Other: Control group received standard therapy

INTERVENTIONS:
Combination Product: extended meropenem infusion in combination with other options such as Polymyxin, Tigecycline, Ertapenem, or Amikacin. — In the case of XDR or PDR Pseudomonas spp. or Acinetobacter spp. isolation from the patient's specimen, treatment was adjusted to extended meropenem infusion in combination with other options such as Polymyxin, Tigecycline, Ertapenem, or Amikacin in group (A) of patients.
  Arms: extended meropenem infusion in combination with other options
Combination Product: two β-lactam antibiotics plus a single non-β-lactam antibiotic — In the case of XDR or PDR Pseudomonas spp. or Acinetobacter spp. isolation from the patient's specimen, treatment was adjusted to include two β-lactam antibiotics plus a single non-β-lactam antibiotic, or a combination of double β-lactam antibiotics, with the aim of avoiding aggressive and toxic antibiotics in group (B) of patients
  Arms: two β-lactam antibiotics plus a single non-β-lactam antibiotic
Other: Control group received standard therapy — Treatment was adjusted to the second-line empirical antibiotic according to the hospital's local policy.
  Arms: c) Patients treatment was adjusted to the second-line empirical antibiotic

SUMMARY:
The goal of this clinical trial is to determine the most effective empirical therapy of antibiotics for better ventilator-associated pneumonia control. The main question it aims to answer is:

• Which is better for clinical response single or combination empiric antibiotic therapies ?

ELIGIBILITY:
Inclusion criteria:

-Patients ranging from one month to twelve years old, who had been undergoing mechanical ventilation for over 48 hours and were diagnosed with Ventillator Associated Pneumonia.

2.1.3. Exclusion criteria:

* Patients with pneumonia prior to mechanical ventilation initiation.
* Patients who had been intubated for more than 24 hours before admission to the PICU, or those transferred from other PICUs and were already receiving antibiotic therapy.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Antimicrobial susceptibility | 7 days
  Antimicrobial susceptibility was assessed through Kirby-Bauer's disc diffusion method (DD), Minimal Inhibitory Concentration (MIC) using the automated VITEK 2 compact system (bioMérieux, France), and the Ameri-Ziaei Double Antibiotic Synergism Test (AZDAST). Interpretation of DD and MIC results followed CLSI guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Intensive Care Unit (PICU) at Cairo University's Faculty of Medicine, Cairo, Egypt